CLINICAL TRIAL: NCT06738407
Title: Doxycycline Prophylaxis for Prevention of Sexually Transmitted Infections Among Adolescent and Young Adult Females in the United States
Brief Title: Doxycycline Prophylaxis for Prevention of Sexually Transmitted Infections
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID)/Division of AIDS (DAIDS) (Unknown); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); Florida State University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); The Office of the Director, National Institutes of Health (NIH) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN173/HPTN 115; UM2HD111076 (NIH); UM2HD111102 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gonorrhea; Chlamydia; Syphilis; Sexually Transmitted Infections (STIs)
Keywords: Sexually Transmitted Infections; STIs; Doxycycline Prophylaxis; Doxycycline
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Syphilis; Sexually Transmitted Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 to (1) on-demand doxyPEP (doxycycline 200 mg as soon as possible and within 72 hours after any condomless oral, vaginal, and/or anal sex), (2) weekly doxycycline (doxycycline 200 mg weekly regardless of sexual activity), or (3) SOC (quarterly STI testing/treatment and sexual health counseling). Participants will complete quarterly study visits over the course of 1 year during which they will receive STI testing (GC, CT, and syphilis), complete surveys, undergo safety monitoring, provide specimens for objective markers of doxycycline adherence and other laboratory assessments, and provide specimens (vaginal and rectal swabs [participant self-collected or staff-collected if the participant prefers]) for future testing, such as microbiome analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- On-demand doxyPEP (Experimental): Participants will take by mouth doxycycline 200 mg as soon as possible and within 72 hours after any condomless oral, vaginal, and/or anal sex in addition to standard of care STI testing/treatment and sexual health counseling.
  Interventions: Drug: Doxycycline hyclate delayed released 200 mg
- Weekly doxycycline (Experimental): Participants will take by mouth doxycycline 200 mg weekly regardless of sexual activity in addition to standard of care STI testing/treatment and sexual health counseling.
  Interventions: Drug: Doxycycline hyclate delayed released 200 mg weekly
- Quarterly STI testing/treatment and sexual health counseling (Other): Participants will be followed per standard of care with quarterly STI testing/treatment and sexual health counseling.
  Interventions: Other: Per standard of care with quarterly STI testing/treatment and sexual health counseling

INTERVENTIONS:
Drug: Doxycycline hyclate delayed released 200 mg — 200 mg of doxycycline taken by mouth as soon as possible and within 72 hours after any condomless oral, vaginal, and/or anal sex along with STI screening and sexual health counseling
  Arms: On-demand doxyPEP
Drug: Doxycycline hyclate delayed released 200 mg weekly — 200 mg of doxycycline taken by mouth weekly regardless of sexual activity along with STI screening and sexual health counseling
  Arms: Weekly doxycycline
Other: Per standard of care with quarterly STI testing/treatment and sexual health counseling — Quarterly STI testing/treatment and sexual health counseling
  Arms: Quarterly STI testing/treatment and sexual health counseling

SUMMARY:
The goal of this open-label, randomized trial is to assess the efficacy of doxycycline prophylaxis in reducing incidences of bacterial sexually transmitted infections (STIs) among adolescent and young adult females while also evaluating acceptability and antimicrobial resistance in order to inform public health policy.

DETAILED DESCRIPTION:
Participants will be randomized to receive on-demand doxycycline post-exposure prophylaxis (doxyPEP), weekly doxycycline, or standard of care (SOC) and will be followed quarterly to assess the impact of doxycycline use on the quarterly incidence of STIs (gonorrhea [GC], chlamydia [CT], and early syphilis), and within the doxycycline arms adherence and acceptability of weekly versus on-demand dosing.

Approximately 760 females will be randomized 1:1:1 to (1) on-demand doxyPEP (doxycycline 200 mg as soon as possible and within 72 hours after any condomless oral, vaginal, and/or anal sex), (2) weekly doxycycline (doxycycline 200 mg weekly regardless of sexual activity), or (3) SOC (quarterly STI testing/treatment and sexual health counseling). Participants will complete quarterly study visits over the course of 1 year during which they will receive STI testing (GC, CT, and syphilis), complete surveys, undergo safety monitoring, provide specimens for objective markers of doxycycline adherence and other laboratory assessments, and provide specimens (vaginal and rectal swabs [participant self-collected or staff-collected if the participant prefers]) for future testing, such as microbiome analysis. Resistance testing will be conducted on Staphylococcus (S.) aureus and Neisseria (N.) gonorrhoeae isolates to evaluate for doxycycline and tetracycline resistance, respectively. Participants will also complete weekly assessments of sexual activity and doxycycline adherence via the HealthMpowerment (HMP) application (app).

ELIGIBILITY:
Inclusion Criteria:

* Age 13-29 years, inclusive;
* Self-reports GC, CT, and/or early syphilis diagnosis in the 12 months prior to screening;
* Self-reports condomless (oral, vaginal, and/or anal) intercourse at least once in the 30 days prior to screening
* Is at least 45 kilograms (99.2 pounds) in weight
* Fluent in English (able to read, speak, and understand English);
* Willing to undergo all required study procedures; and
* Willing to provide written informed consent to participate in the study.

Exclusion Criteria:

* Is male;
* Is pregnant, breastfeeding, or planning to become pregnant in the next 12 months;
* Documented history of tetracycline allergy or self-reports an allergy to tetracyclines;
* Current or anticipated use of a medication (e.g., barbiturates, phenytoin, lithium, carbamazepine, systemic retinoids, warfarin) with a contraindicated interaction to doxycycline ;
* Current or planned use of doxycycline for a prolonged period (> 2 weeks) in the 30 days prior to enrollment, including current prescription for doxycycline for STI prophylaxis;
* Prolonged antibiotic use (> 2 weeks) within the last 30 days prior to enrollment;
* Co-enrollment in any other concurrent interventional research or studies that may interfere with this study, such as an STI prevention trial, unless approved by Protocol Team in writing;
* Does not have consistent access (or anticipated weekly access for 52 weeks of survey completion) to smartphone that can access the HMP app; or
* Any other medical condition, medical/behavioral intervention, or other conditions that, in the opinion of the clinical site Project Lead (PL)/Investigator of Record (IoR) or designee, could interfere with adherence to study procedures or compromise interpretation of study results.

Ages: 13 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 760 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Combined incidence of GC, CT, and/or early syphilis infection | One (1) year
  Overall combined incidence of GC, CT, and/or early syphilis infection by laboratory-based diagnosis (defined as positive GC or CT on nucleic acid amplification test [NAAT] or first positive rapid plasma reagin [RPR] with positive treponemal-specific antibody [Ab] or a new 4-fold rise in RPR titers) over the duration of follow-up.

SECONDARY OUTCOMES:
Individual incidence diagnoses of GC, CT, and early syphilis infection | One (1) year
  Individual incidence diagnoses of GC, CT, and early syphilis infection by laboratory-based diagnosis (defined as positive GC or CT on NAAT or first positive RPR with positive treponemal-specific Ab or a new 4-fold rise in RPR titers) per quarter, by arm.

OTHER OUTCOMES:
First occurrence of a bacterial STI | One (1) year
  First occurrence of a bacterial STI (GC, CT, and/or early syphilis) after study enrollment, based on testing during each quarterly follow-up visit or documented testing occurring at an outside clinical site, by arm.
Proportion GC isolates that are detected as tetracycline-resistant | One (1) year
  Proportion of GC isolates that are detected as tetracycline-resistant during follow-up, by arm.
Proportion S. aureus isolates that are detected as doxycycline-resistant | One (1) year
  Proportion of S. aureus isolates that are detected as doxycycline-resistant at 24 and 48 weeks, by arm.
Adherence to doxycycline | One (1) year
  Adherence to on-demand doxyPEP and weekly doxycycline assessed with objective doxycycline plasma, and/or DBS concentrations matched with expected detection of once-weekly dosing or based on self-reported sexual behavior, by arm.
Adherence to doxycycline - self report | 1 year
  Adherence to on-demand doxyPEP and weekly doxycycline assessed with self- reported proportion of sexual exposures within the prior 12 weeks when on-demand doxyPEP and weekly doxycycline was used, by arm.
Acceptability and optimism | One (1) year
  Acceptability and optimism, using Likert scales, by arm.

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Blaire, MD, PhD, Study Chair — University of California, Los Angeles; Jenell Stewart, DO, MPH, Study Chair — Hennepin Healthcare
Locations (12):
- United States (12):
  - UCLA Care, Los Angeles, California
  - San Francisco Department of Public Health, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Tampa, Florida
  - Ponce de Leon, Atlanta, Georgia
  - University Illinois Chicago, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - Harlem Prevention Center, New York, New York
  - Chapel Hill, Chapel Hill, North Carolina
  - Penn Prevention, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No